CLINICAL TRIAL: NCT01843465
Title: Improving the Assessment of Pulmonary Vein Disconnection With the Achieve Catheter During Atrial Fibrillation Cryoablation
Brief Title: Cryoablation of AF: Improving the Use of the Achieve Catheter
Status: Completed | Type: Observational
Sponsor: Clinique Pasteur (Other)
Responsible Party: Principal Investigator, Serge Boveda, M.D., Clinique Pasteur
Other Study IDs: CP-CRYO-001
Record Dates: First submitted 2013-04-26; First posted 2013-04-30 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-10

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; balloon cryoablation; pulmonary veins
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cryoablation of atrial fibrillation
  Interventions: Other: Maneuvers for documenting the disconnection

INTERVENTIONS:
Other: Maneuvers for documenting the disconnection
  Other Names: type 1; type 2; type 3; type 4

SUMMARY:
According to data from high volume Centres, documentation of entry block with the Achieve catheter may be possible in only about to 50% of pulmonary veins. The investigators aim to assess strategies using the Achieve catheter that can improve this performance.

ELIGIBILITY:
Inclusion Criteria:

* all consecutive patients undergoing atrial fibrillation cryoballoon ablation monitored with the Achieve catheter.

Exclusion Criteria:

* patients in AF at the beginning of the procedure
* patients with a previous AF ablation procedure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients undergoing cryoablation of atrial fibrillation using the Achieve catheter to document pulmonary vein disconnection.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2013-04; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Serge Boveda, M.D., Principal Investigator — Clinique Pasteur
Locations (1):
- Clinique Pasteur, Toulouse, Haute-Garonne, France

REFERENCES:
- [Derived] Boveda S, Providencia R, Albenque JP, Combes N, Combes S, Hireche H, Casteigt B, Bouzeman A, Jourda F, Narayanan K, Marijon E. Real-time assessment of pulmonary vein disconnection during cryoablation of atrial fibrillation: can it be 'achieved' in almost all cases? Europace. 2014 Jun;16(6):826-33. doi: 10.1093/europace/eut366. Epub 2013 Dec 18. PMID 24351882

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were recruited at Clinique Pasteur. During the inclusion period, 36 underwent cryoballoon ablation of atrial fibrillation using the Achieve 20mm catheter for real-time documentation of PV potentials.
Pre-assignment Details: 2 patients were not considered eligible due to previous atrial fibrillation ablation.
Groups:
- Cryoablation of Atrial Fibrillation: All patients underwent cryoballoon ablation of atrial fibrillation using the Achieve 20mm catheter for real-time documentation of PV potentials.
  According to the maneuvers for documenting the disconnection , 4 PV types were defined:
  Type 1 - Achieve allowing documentation of PV disconnection in the standard position.
  Type 2 - Need of backward/proximal displacement of the Achieve catheter to display PV potentials during cryoenergy application.
  Type 3 - No possibility of clear documentation of PV potentials, but capture of PV with pacing Type 4 - no real-time documentation of PV disconnection
Period: Overall Study
Arm/Group | Cryoablation of Atrial Fibrillation
Started | 34 (This study had no follow-up. It focused in the acute setting of cryoballoon ablation.)
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Cryoablation of Atrial Fibrillation: Maneuvers for documenting the disconnection :
Arm/Group | Cryoablation of Atrial Fibrillation
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 59.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 21
Region of Enrollment [Number; unit: participants]
  France | 34

OUTCOME MEASURES:

1. Primary Outcome: Real-time Documentation of Pulmonary Vein Disconnection
Description: Possibility of real-time documentation of the pulmonary vein during cryoballoon ablation, through the use of the Achieve catheter. This will be codified as "yes" or "no", and in case of an affirmative answer Final results will be expressed as a % of the total pulmonary veins where disconnection was documented in real-time and the time of maneuver of the Achieve catheter that was necessary i.e. standard position (type 1); withdrawal position (type 2) or need of pacing (type 3). A pulmonary vein where no real-time documentation is possible, will be named as a type 4.
Time Frame: atrial fibrillation cryoablation procedure
Population: According to the different pulmonary vein anatomies in the study sample, 128 pulmonary veins were assessed.
Measure: Number; unit: number of PVs disconnected in realtime
Units Other Than Participants: pulmonary veins
Groups:
- Cryoablation of Atrial Fibrillation: Maneuvers for documenting the disconnection :
  Type 1 pulmonary veins Type 2 pulmonary veins Type 3 pulmonary veins Type 4 pulmonary veins
Arm/Group | Cryoablation of Atrial Fibrillation
Number analyzed (Participants) | 34
Number analyzed (pulmonary veins) | 128
number of PVs disconnected in realtime | 125

ADVERSE EVENTS:
Arm/Group | Cryoablation of Atrial Fibrillation
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 2/34
OTHER ADVERSE EVENTS (reported when occurring in more than 2.9% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cryoablation of Atrial Fibrillation (N=34)
phrenic nerve palsy lasting > 24 hours (Musculoskeletal and connective tissue disorders) | 1 (1)
atrial fibrillation of left atrial flutter recurrence in the first 24 hours (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes